CLINICAL TRIAL: NCT03689959
Title: Correction of Fixed Knee Flexion Deformity in Children Using Eight-plate Hemiepiphysiodesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Yahya Abdel Azeem Hassanein, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMIN000018950
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Knee Deformity
Keywords: knee; flexion deformity; hemiepiphysiodesis; eight plate; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): 13 child with fixed knee flexion deformity more than 10° on one or both sides with 12 months or more predicted growth remaining subjected to eight plate hemiepiphysiodesis of the distal femur
  Interventions: Procedure: Eight plate hemiepiphysiodesis

INTERVENTIONS:
Procedure: Eight plate hemiepiphysiodesis — Patient is positioned in a classic supine position. Under fluoroscopic guidance and tourniquet hemostasis, the distal femoral physis is identified. Two 3-cm incisions are made, one on either side of the patella, centred at the level of the physis. The capsule and synovium are opened to visualize the sulcus and place the plates just outside the articular portion of the joint surface, medially and laterally. Care is taken not to damage the periosteum and a needle is inserted into the physis. The 8-plate, which has a central hole, is slipped over the needle and screws inserted. After wound closure, a soft dressing is used, and the patient is allowed to ambulate as tolerated.
  Other Names: Guided growth

SUMMARY:
The study aims to assess the effectiveness of hemiephysiodesis using eight plates in correction of fixed knee flexion deformities in children.

DETAILED DESCRIPTION:
Flexion contractures of the knee are quite disabling. They produce deleterious effects on knee biomechanics, quadriceps function, energy expenditure during gait and the overall ability to ambulate. These deformities occur secondary to a number of different etiologies including; congenital, traumatic, inflammatory and neuromuscular disorders with cerebral palsy (CP) being on the top of the list.

The main aim of correction of sagittal plane deformities of the knee is to restore the range of motion. Surgical options available for correction of knee flexion contractures include soft tissue modification, acute correction by osteotomies, gradual correction by external fixators and growth modulation by hemiephysiodesis.Extensive soft tissue surgery may be needed for correction of knee deformities with potential risk of neurovascular damage and wound complications. Supracondylar extension osteotomies have been widely used, however prolonged immobilization and associated neurovascular insults have always been major concerns. External fixators are cumbersome and may produce muscle tethering and pin tract infections.

There are few studies in the literature reporting the use of anterior hemiepiphysiodesis for correction of knee flexion contracture.

Our study question can be summarized as follows; Is hemiepiphysiodesis by eight plates effective for correction of fixed knee flexion deformities in children ?

ELIGIBILITY:
Inclusion Criteria:

* Fixed knee flexion deformity more than 10°
* Unilateral or bilateral cases
* 12 months or more predicted growth remaining
* No response to non-operative treatment (physical therapy, bracing, casting);
* Recurrent cases

Exclusion Criteria:

* Dynamic deformities due to spasticity
* Deformities responding to conservative treatment

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Degree of flexion deformity | One year
  The angle between the anterior borders of thigh and leg measured clinically with a goniometer

SECONDARY OUTCOMES:
Complications | One year
  Wound complications, metal failure
Rate of correction | One year
  Time needed for correction of deformity

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y. Hassanein, M.Sc., Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Spiro AS, Stenger P, Hoffmann M, Vettorazzi E, Babin K, Lipovac S, Kolb JP, Novo de Oliveira A, Rueger JM, Stuecker R. Treatment of fixed knee flexion deformity by anterior distal femoral stapling. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2413-8. doi: 10.1007/s00167-012-1915-8. Epub 2012 Feb 4. PMID 22307752
- [Result] Klatt J, Stevens PM. Guided growth for fixed knee flexion deformity. J Pediatr Orthop. 2008 Sep;28(6):626-31. doi: 10.1097/BPO.0b013e318183d573. PMID 18724198
- [Result] Spiro AS, Babin K, Lipovac S, Rupprecht M, Meenen NM, Rueger JM, Stuecker R. Anterior femoral epiphysiodesis for the treatment of fixed knee flexion deformity in spina bifida patients. J Pediatr Orthop. 2010 Dec;30(8):858-62. doi: 10.1097/BPO.0b013e3181f10297. PMID 21102213
- [Result] Heydarian K, Akbarnia BA, Jabalameli M, Tabador K. Posterior capsulotomy for the treatment of severe flexion contractures of the knee. J Pediatr Orthop. 1984 Nov;4(6):700-4. doi: 10.1097/01241398-198411000-00009. PMID 6511897
- [Result] Inan M, Sarikaya IA, Yildirim E, Guven MF. Neurological complications after supracondylar femoral osteotomy in cerebral palsy. J Pediatr Orthop. 2015 Apr-May;35(3):290-5. doi: 10.1097/BPO.0000000000000264. PMID 25075896
- [Result] Carbonell PG, Valero JV, Fernandez PD, Vicente-Franqueira JR. Monolateral external fixation for the progressive correction of neurological spastic knee flexion contracture in children. Strategies Trauma Limb Reconstr. 2007 Dec;2(2-3):91-7. doi: 10.1007/s11751-007-0026-4. Epub 2007 Dec 4. PMID 18427750